CLINICAL TRIAL: NCT02915692
Title: A Clinical Study to Compare the CAUTI Rates Following ERASE CAUTI Tray Silver Coated Foley Catheters Verse Silver Coated Foley Catheters
Brief Title: Study to Compare CAUTI Rates Following ERASE CAUTI Tray Silver vs Silver Coated Foley Catheters
Status: Terminated | Type: Observational
Why Stopped: Withdrawn funding
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Other Study IDs: MII-002
Record Dates: First submitted 2012-02-09; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Surgery
Keywords: Foley; CAUTI; ERASE CAUTI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ERASE Silver Coated Foley Catheters: Subjects given silver catheters from an ERASE CAUTI Tray.
  Interventions: Device: ERASE Silver Coated Foley Catheter
- Comparator Silver Coated Catheter: Comparator silver urinary catheter
  Interventions: Device: Comparator Silver Coated Catheter

INTERVENTIONS:
Device: ERASE Silver Coated Foley Catheter — Foley catheter from ERASE CAUTI Kit will be administered as required.
  Other Names: Silver coated Foley catheter
  Groups: ERASE Silver Coated Foley Catheters
Device: Comparator Silver Coated Catheter — Foley catheter coated with silver
  Other Names: Silver coated catheter
  Groups: Comparator Silver Coated Catheter

SUMMARY:
The Foley catheter is one component in a catheter insertion procedure that could contribute to a catheter associated urinary tract infection (CAUTI). Improvements in the catheter insertion procedure using the ERASE CAUTI Tray system may help to lower these infection rates.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Received either silver coated Foley catheter or ERASE CAUTI silver coated catheter

Exclusion Criteria:

* UTI present upon current hospital admission
* Burn patients, transplant patients, or immune-compromised patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring Foley catheters
Sampling Method: Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection rates | 2 days on average or until hospital discharge
  Infection rate/1000 catheter days based on days of use. As the number of days a catheter is used varies, the minimum expected time frame on average is 2 days. However, infections will be monitored during catheter use.

SECONDARY OUTCOMES:
Catheter use | 2 days on average or until hospital discharge
  The average number of days a catheter is used is typically 2 days. However during the hospital stay, the time a catheter remains varies on medical need. The total daily use of each catheter will be tabulated after removal..
Catheter Associated Urinary Track Infection Costs | Post Infection costs incurred from insertion of catheter to hospital discharge (<30 days)
  Costs associated with urinary track Infections during the use of a catheter in the study will calculated from the time infection was identified until hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: S T Symeonides, MD, Principal Investigator — Parish Medical Center
Locations (1):
- Oconnee Regional Medical Center, Milledgenville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No